CLINICAL TRIAL: NCT06390267
Title: Effect of Transcutaneous Auricular Neurostimulation on Cognitive Performance in a Laboratory Model of Acute Stress Reaction
Acronym: ASR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Biomedical, Inc. (Industry)
Collaborators: Battelle Memorial Institute (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBM-ASR-01
Record Dates: First submitted 2024-04-17; First posted 2024-04-30 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Acute Stress Reaction; Cognitive Performance
Keywords: Healthy Human; Performance; Stress; Vagus Nerve Stimulation; Neurostimulation; Transcutaneous Auricular Neurostimulation; Military
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized, double-blind, sham-controlled trial in sixty healthy, able-bodied participants. Participants will be randomized to one of four treatment groups in a 1:1:2:2 ratio. Twice as many participants will be randomized to the acute treatment active tAN and acute treatment sham tAN arms (Groups 3 and 4) compared to the prophylactic treatment group arms (Groups 1 and 2).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study investigators and personnel delivering assessments will be blind to whether patient is assigned to an active or sham tAN group. This will ensure a non-biased assessment of post-stressor performance. All participants will be blinded to whether they are receiving active or sham tAN. Participants will complete a blinding effectiveness questionnaire at the conclusion of the study. To maintain the blind, all participants will be informed that "you may or may not perceive stimulation, meaning you may receive benefits without any perception of stimulation."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Active tAN for Prophylactic Treatment (Experimental): Prophylactic Active participants will undergo 20 minutes of active tAN while remaining seated and idle. After stimulation, participants will proceed into the 20-minute stressor protocol.
  Interventions: Device: Sparrow Hawk (Active)
- Sham Stimulation for Prophylactic Treatment (Sham Comparator): Prophylactic Sham participants will undergo 20 minutes of sham stimulation while remaining seated and idle. After stimulation, participants will proceed into the 20-minute stressor protocol.
  Interventions: Device: Sparrow Hawk (Sham)
- Active tAN for Acute Treatment (Experimental): Acute Active participants will begin the stressor protocol immediately after baseline assessments. After a 5-min period of the stressor protocol without any intervention, active tAN treatment will be delivered concurrently for the remainder of the stressor protocol for a total of 20 minutes of stimulation and approximately 25 minutes of the stressor protocol.
  Interventions: Device: Sparrow Hawk (Active)
- Sham Stimulation for Acute Treatment (Sham Comparator): Acute Sham participants will begin the stressor protocol immediately after baseline assessments. After a 5-min period of the stressor protocol without any intervention, sham stimulation will be delivered concurrently for the remainder of the stressor protocol for a total of 20 minutes of stimulation and approximately 25 minutes of the stressor protocol.
  Interventions: Device: Sparrow Hawk (Sham)

INTERVENTIONS:
Device: Sparrow Hawk (Active) — Wearable, battery-operated, device designed to transcutaneously stimulate nerves on and/or around the auricle. The device will be used to deliver tAN sessions of active (prophylactic or acute) therapy according to the participant's randomization group.
  Arms: Active tAN for Acute Treatment; Active tAN for Prophylactic Treatment
Device: Sparrow Hawk (Sham) — Wearable, battery-operated, device designed to transcutaneously stimulate nerves on and/or around the auricle. The device will be used to deliver tAN sessions of sham (prophylactic or acute) therapy according to the participant's randomization group.
  Arms: Sham Stimulation for Acute Treatment; Sham Stimulation for Prophylactic Treatment

SUMMARY:
The objective of this study is to test the effects of transcutaneous auricular neurostimulation (tAN) in treating or preventing performance degradation after an acute stressor.

DETAILED DESCRIPTION:
This study is designed as a randomized, double-blind, sham-controlled trial. Sixty healthy, able-bodied participants will be randomized 1:1:2:2 into one of four experimental groups:

Group 1: Active tAN for prophylactic treatment prior to acute stress exposure (N=10)

Group 2: Sham stimulation for prophylactic treatment prior to acute stress exposure (N=10)

Group 3: Active tAN for acute treatment during acute stress exposure (N=20)

Group 4: Sham stimulation for acute treatment during acute stress exposure (N=20)

Participants will complete a baseline performance of three tasks. tAN treatment will then be administered prior to or during an acute stress test. Participants will complete the same three tasks preformed at baseline. In addition to the tAN therapy earpiece, subjects will have biosensors attached to them to collect biomarker information.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 41 years old
2. Participant has the cognitive and physical abilities to carry out the study tasks
3. Proficient in the English language
4. Ability to understand the explanations and instructions given by the study personnel

Exclusion Criteria:

1. Participant presents current evidence of an uncontrolled and/or clinically significant medical condition or psychiatric condition
2. Participant has used any psychological stress-management intervention within the last 4 weeks
3. Participant is participating in another interventional trial within 90 days prior to or throughout duration of trial
4. Participant has a prior diagnosis of post-traumatic stress disorder, acute stress disorder, or generalized anxiety disorder
5. Participant is currently using anti-anxiety medications such as Xanax or beta blockers
6. Participant has a diagnosis of attention deficit hyperactivity disorder (ADHD) and/or is currently taking medications for the treatment of ADHD.
7. History of substance abuse or drug dependence including nicotine and alcohol in the past 3 months
8. Participant has abnormal ear anatomy, ear infection present, or earpiercing that could interfere with stimulation
9. Participant has a history of epileptic seizures
10. Participant has a history of neurologic diseases or traumatic brain injury
11. Participant wears or utilized other devices that cannot be removed during the study (e.g., pacemakers, cochlear prostheses, neurostimulators)
12. Females who are pregnant or lactating
13. Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants are risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Match-to-Sample Task (MST) | From baseline to post-stressor (up to 3 hours)
  Mean change in performance on the MST (in combination with the Psychomotor Vigilance Task (PVT) and Perdue Pegboard Task (PPT)) in the active tAN acute treatment group (Group 3) compared to sham acute treatment group (Group 4). The MST assesses short-term spatial memory (working memory) and pattern recognition skills. An 8 × 8 matrix of a red and green checkerboard pattern will be presented for 10 seconds, then removed, and then followed by a variable delay of 8 or 16 seconds. Two matrices will then be presented: the original matrix and a matrix with the color of 2 squares reversed. The subjects will attempt to select the original matrix. The task consists of 30 trials, ≈15 for each delay. A response (left or right arrow key) is required within 10 s, or a time-out error will be recorded. Correct matches were recorded, as was reaction time. This test takes less than 5 minutes to complete.
Psychomotor Vigilance Task (PVT) | From baseline to post-stressor (up to 3 hours)
  Mean change in performance on the PVT (in combination with the MST and PPT) in the active tAN acute treatment group (Group 3) compared to sham acute treatment group (Group 4). The PVT is a test of visual reaction time. A series of stimuli are presented at random intervals on a screen, and the subject responds as rapidly as possible when a stimulus appears. Response time, false alarms, and the number of lapses (long duration responses) will be recorded. Performance lapses refer to the instances when a subject failed to respond in <500 ms. This test will be administered on a computer monitor or tablet.
Perdue Pegboard Task (PPT) | From baseline to post-stressor (up to 3 hours)
  Mean change in performance on the PTT (in combination with the PVT and MST) in the active tAN acute treatment group (Group 3) compared to sham acute treatment group (Group 4). The PPT is a psychomotor test of manual dexterity and bimanual coordination. A pegboard consisting of two parallel sets of twenty-five holes arranged vertically is presented to the participant, and they are asked to remove pegs from concave cups at the top of the board and place them in the holes sequentially as rapidly as possible. The number of pegs placed successfully in thirty seconds is scored. Each participant is tested three times using both hands.
Maastricht Acute Stress Test (MAST) | After baseline tasks, approximately 35 minutes
  The MAST is a safe, non-invasive, and expedited method to create a stress response in human subjects under laboratory conditions. The test combines two well-validated laboratory stress paradigms, the Trier Social Stress Test (TSST) and the Cold Pressor Test (CPT) into a single protocol. The MAST is effective in increasing salivary cortisol, increasing blood pressure, salivary alpha-amylase, and eliciting subjective stress reactions. Participants will be videotaped and monitored to analyze their facial expressions. They will undergo multiple hand immersion trials (HIT) in which they have to immerse their hand in ice-cold (2 °C) water. They will engage in mental arithmetic trials (MAT), counting backwards starting at 2043 in steps of 17 as fast and accurate as possible. For each mistake made, the experimenter will provide negative feedback and instruct them to start over at 2043.

SECONDARY OUTCOMES:
Mean change in performance on the MST in the active tAN groups (Groups 1 and 3) compared to sham groups (Groups 2 and 4). | From baseline to post-stressor (up to 3 hours)
  Mean change in performance on the MST in combination with PVT and PPT
Mean change in performance on the PVT in the active tAN groups (Groups 1 and 3) compared to sham groups (Groups 2 and 4). | From baseline to post-stressor (up to 3 hours)
  Mean change in performance on the PVT in combination with MST and PPT
Mean change in performance on the PPT in the active tAN groups (Groups 1 and 3) compared to sham groups (Groups 2 and 4). | From baseline to post-stressor (up to 3 hours)
  Mean change in performance on the PPT in combination with MST and PVT
Mean change in performance on the MTS in the prophylactic active tAN group (Group 1) compared to the acute active tAN group (Group 3). | From baseline to post-stressor (up to 3 hours)
  Mean change in performance on the MST in combination with PVT and PPT
Mean change in performance on the PVT in the prophylactic active tAN group (Group 1) compared to the acute active tAN group (Group 3). | From baseline to post-stressor (up to 3 hours)
  Mean change in performance on the PVT in combination with MST and PPT
Mean change in performance on the PPT in the prophylactic active tAN group (Group 1) compared to the acute active tAN group (Group 3). | From baseline to post-stressor (up to 3 hours)
  Mean change in performance on the PPT in combination with MST and PVT
Change in working memory as measured by performance on the MST | From baseline to post-stressor (up to 3 hours)
Change in reaction time as measured by performance on the PVT | From baseline to post-stressor (up to 3 hours)
Change in dexterity as measured by performance on the PPT | From baseline to post-stressor (up to 3 hours)

OTHER OUTCOMES:
Change in heart rate variability in milliseconds (ms) across groups | From baseline, during the stressor, and post-stressor (up to 3 hours)
  Biomarker data will be collected throughout the study using wearable sensors, including the off-the-shelf Empatica E4 smart watch and the Corti SweatSensor.
Change in heart rate in beats per minute (bpm) across groups | From baseline, during the stressor, and post-stressor (up to 3 hours)
  Biomarker data will be collected throughout the study using wearable sensors, including the off-the-shelf Empatica E4 smart watch and the Corti SweatSensor.
Change in electrodermal activity across groups | From baseline, during the stressor, and post-stressor (up to 3 hours)
  Biomarker data will be collected throughout the study using wearable sensors, including the off-the-shelf Empatica E4 smart watch and the Corti SweatSensor.
Change in cortisol levels across groups | From baseline, during the stressor, and post-stressor (up to 3 hours)
  Biomarker data will be collected throughout the study using wearable sensors, including the off-the-shelf Empatica E4 smart watch and the Corti SweatSensor.
Change in Interleukin-6 (IL-6) levels across groups | From baseline, during the stressor, and post-stressor (up to 3 hours)
  Biomarker data will be collected throughout the study using wearable sensors, including the off-the-shelf Empatica E4 smart watch and the Corti SweatSensor.
Change in melatonin levels across groups | From baseline, during the stressor, and post-stressor (up to 3 hours)
  Biomarker data will be collected throughout the study using wearable sensors, including the off-the-shelf Empatica E4 smart watch and the Corti SweatSensor.
Change in Tumor Necrosis Factor Alpha (TNF-α) levels across groups | From baseline, during the stressor, and post-stressor (up to 3 hours)
  Biomarker data will be collected throughout the study using wearable sensors, including the off-the-shelf Empatica E4 smart watch and the Corti SweatSensor.
Change in self-reported stress across groups using the Stress Monitoring and Response Tool (SMART) | Before baseline to after post-stressor tasks (up to 3 hours; assessment valid up to 24 hours after event))
  The SMART tool is a patient-reported assessment of acute stress. The questionnaire contains questions asking the participant to rate their severity of stress related symptoms on a scale of 0 ("none") to 10 ("severe"). Symptoms include feeling worthless, sad, distant, irritable, headaches, dizziness, fatigue, nausea, difficulty concentrating, pain, etc. This study will ask participants 23 questions on the SMART tool based on their recent experiences.
Mean therapeutic stimulation intensity | From start to end of tAN (30 minutes)
  amplitude in milliamperes (mA)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Putnam, PhD, Principal Investigator — Battelle Memorial Institute; Navid Khodaparast, PhD, Principal Investigator — Spark Biomedical, Inc.
Locations (1):
- Battelle Memorial Institute, Columbus, Ohio, United States